CLINICAL TRIAL: NCT02300012
Title: A Pilot Study to Investigate Biomarkers in ACL Patients and Healthy Controls
Brief Title: A Pilot Study to Investigate Biomarkers in Anterior Cruciate Ligament (ACL) Patients and Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Lincolnshire Hospitals NHS Trust (Other)
Collaborators: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 120614Mullineaux
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior cruciate ligament; Performance based investigations
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Operation - No PBI (No Intervention): Patients requiring operation - baseline PBI data not seen by surgeon
- Operation - PBI available (Experimental): Patients requiring operation - baseline PBI data seen by surgeon pre-operatively
  Interventions: Procedure: Surgeons knowledge of pre-operative PBIs
- Non-operation (No Intervention): Patients with ACL rupture not requiring operation
- Control (No Intervention): Healthy age matched volunteers - No operation

INTERVENTIONS:
Procedure: Surgeons knowledge of pre-operative PBIs — Surgeon performing ACL repair will have prior knowledge of patients pre-operative PBIs to inform surgical practice
  Arms: Operation - PBI available

SUMMARY:
Incident rates of ACL rupture are greatest in 16-39 year olds at almost 1 in 1,000.

Performance Based Investigations (PBIs) can be used to evaluate and select correct approaches to patient treatment, and biochemical, biomechanical and physiological biomarkers in other conditions are sensitive in distinguishing between disease state severities, type of injuries and responsiveness to treatment. Despite the measurement sensitivity of PBIs, these are not widely used possibly owing to their focus postoperatively where benefits are less worthwhile.

This study aims to investigate novel biomarkers as performance based investigations (PBIs) to improve surgical and treatment strategies in anterior cruciate ligament (ACL) patients. The objectives are to identify whether biomarkers, collected before and after operations, can: 1) Assist the surgeon in decision making; 2) Lead to improved prognosis; 3) Be used to predict the outcomes of prognosis, and; 4) Correlate with disease signs/ smoking to help further understand ACL injuries.

ELIGIBILITY:
Inclusion Criteria:

* unilateral ACL rupture
* 18 - 45 years old

Exclusion Criteria:

* combined posterior and ACL rupture
* multi-ligament instability including medial or lateral collateral ligament injury
* other lower limb surgery <3mths
* current significant acute injury affecting other lower extremity joints, or other relevant neurological or musculoskeletal pathology.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
The change in knee varus/valgus from baseline to 6 weeks post-ACL reconstruction, measured when performing a single leg squat. | Baseline, 6 weeks
The change in knee varus/valgus from baseline to 6 months post-ACL reconstruction, measured when performing a single leg squat | Baseline, 6 months
The change in peak vertical ground reaction force from baseline to 6 weeks post-ACL reconstruction, measured when performing a novel isometric task during sitting. | Baseline, 6 weeks
The change in peak vertical ground reaction force from baseline to 6 months post-ACL reconstruction, measured when performing a novel isometric task during sitting. | Baseline, 6 months
The change in anterior-posterior centre of pressure displacement from baseline to 6 weeks post-ACL reconstruction, measured when performing a 10 second standing balance task. | Baseline, 6 weeks
The change in anterior-posterior centre of pressure displacement from baseline to 6 months post-ACL reconstruction, measured when performing a 10 second standing balance task. | Baseline, 6 months
The change in time taken to complete a sit-to-stand task, from baseline to 6 weeks post-ACL reconstruction | Baseline, 6 weeks
The change in time taken to complete a sit-to-stand task, from baseline to 6 months post-ACL reconstruction | Baseline, 6 months

SECONDARY OUTCOMES:
The change in Interleukin-6 obtained from blood samples at baseline to 6 months post-ACL reconstruction | 6 months post-ACL reconstruction
The change in Tegner Activity Score from baseline to 6 months post-ACL reconstruction | 6 months post-ACL reconstruction
The change in Lysholm Knee Scoring Scale from baseline to 6 months post-ACL reconstruction | 6 months post-ACL reconstruction
The change in International Knee Documentation Committee subjective knee evaluation form from baseline to 6 months post-ACL reconstruction | baseline to 6 months post-ACL reconstruction
The difference in bone morphogenetic protein-7 (BMP-7) between smokers and non-smokers who undergo ACL reconstruction | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Prof David Mullineaux, PhD, Principal Investigator — University of Lincoln
Locations (1):
- United Lincolnshire Hospitals NHS Trust, Lincoln, Lincolnshire, United Kingdom